CLINICAL TRIAL: NCT04753450
Title: Correlation of Muscle Ultrasound Measures (2D and 3D) With Biphotonic X-ray Absorptiometry in Oldest Old Patients.
Acronym: DIASEM
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC20_0534
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Assessment, Self; Muscle Atrophy; Ultrasound Therapy; Complications; Aging
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The sarcopenia diagnosis is based on the muscle mass and on impaired physical performance. The emerging field of ultrasound assessment of muscle mass in older patients is based on 2d parameters with prediction equations for muscle mass. For the moment, validation of prediction equations in older adults with varying function and health is lacking. The study aims to evaluate correlation of muscle mass between 3D muscle mass measurement and DXA, in order to dispense with the prediction equation.

DETAILED DESCRIPTION:
Older patients who agree to participate to the study will undergo 3D ultrasound muscle mass measurement, 2D panoramic mode muscle mass measurement and biphotonic X-ray absorptiometry assessment. Correlation analysis will be done with the different measurement.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 75 years old
* Osteoporosis diagnosis confirmed by Dual-energy X-ray Absorptiometry

Exclusion Criteria:

* Neurocognitive disorders preventing the expression of informed consent
* Patients who cannot undergo an examination in a static position
* Lack of a measurement site (muscle resection or amputation)
* Any state of dehydration or water inflation
* Patient with legal protection measure

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older patients who agrees to participate to the study will undergo 3D ultrasound muscle mass measurement, 2D panoramic mode muscle mass measurement and biphotonic X-ray absorptiometry assessment, the same day. Correlation analysis will be done with the different measurement.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
3D Correlation between muscle volume measured by 3D ultrasound and standard method : DXA results | 1 week
  Correlation between muscle volume measured by 3D ultrasound and standard method : DXA results

SECONDARY OUTCOMES:
2D correlation between muscle volume measured by 2D ultrasound and standard method : DXA results | 1 week
  Correlation between muscle volume measured by 2D ultrasound and standard method : DXA results

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided